CLINICAL TRIAL: NCT04492215
Title: Improving the Participation Rate in ColoRectal Cancer Screening by Training General Practitioners in Motivational Interviewing
Brief Title: General Practitioners and Participation Rate in ColoRectal Cancer Screening
Acronym: AMDepCCR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 29BRC19.0115 (AMDepCCR); 2019-A01776-51 (Other: IDRCB)
Record Dates: First submitted 2020-07-27; First posted 2020-07-30 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-04

CONDITIONS: Colorectal Cancer
Keywords: Colorectal cancer; General practitioners; Motivational interviewing
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Motivational Interviewing

STUDY DESIGN:
Intervention Model Description: This study is a multicenter trial. Patients will be followed either by GPs from the interventional group who participated in motivational interviewing or by the control group who never participated. The distribution of general practitioners in the groups is done thanks random draw.
Who Masked: Participant
Masking Description: The study is based on the participation of general practitioners in a training, the test is necessarily open for doctors. However patients will not know if their doctor has received training and will be blinded..
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physicians trained in motivational interviewing (Experimental): Patients followed by general practitioners trained in motivational interviewing
  Interventions: Behavioral: Interaction between patient and trained general practitioners in motivational interviewing
- Physicians did not trainned in motivational interviewing (No Intervention): Patients followed by general practitioners who did not receive motivational interviewing.

INTERVENTIONS:
Behavioral: Interaction between patient and trained general practitioners in motivational interviewing — Impact of the medical interview on the patient
  Other Names: Experimental arm
  Arms: Physicians trained in motivational interviewing

SUMMARY:
Colorectal cancer is the 2nd leading cause of cancer mortality in France. However this cancer is preventable in the majority of cases by early detection of adenomas.

In France, there is organized colorectal cancer screening, which relies on general practitioners (GPs). Tests delivered by GPs are performed in 89% of cases. However, GPs do not systematically offer the test, for time management and communication reasons. Patients expect their GPs to offer the test and to focus on their expectations. A previous study conducted on GPs showed that training in communication and motivational interviewing increases the number of tests performed by 12.2%.

In order to facilitate the promotion of screening, the investigators would like to develop a training programme for GPs focusing on the application of Motivational Interviewing (MI) techniques to the promotion of colorectal cancer screening.

Motivational Interviewing is a directive, client-centered counseling style for eliciting behavior change by helping clients to explore and resolve ambivalence.

This study is a multicenter trial in general medicine. In this randomized trial the 902 subjects will be included prospectively by the general practitioners (GP) participating in the study.

As a first step, general practitioners who have never participated in Motivational Interviewing training will be recruited and split into 2 groups by randomization, an intervention group and a control group. The interventional group will then undergo a 3 times 2-day training in Motivational Interviewing.

In a second step, the patients will be included by those GP and a self-questionnaire will be send at the inclusion and after 6, 12 and 24 months. The evaluation of the number of tests performed and the analyse of the Health Belief Model (HBM) self-questionnaire will be carried out.

At 24 months, there will be an evaluation of the denial motivation questionnaire for patients who have not participated in organized colorectal cancer screening.

ELIGIBILITY:
Inclusion Criteria:

* People with an average risk of colorectal cancer (presenting no symptoms or risk factors).
* People living in Finistère.
* People aged 50 to 74 who have never participated in organized screening for colorectal cancer.

Exclusion Criteria:

* Persons without address to receive the Health Belief Model (HBM)questionnaire
* People who do not fit the organized screening criteria
* Persons unable to give consent (patients under guardianship, curatorship, non-French speaking, illiterate)

Ages: 50 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 902 (Estimated)
Dates: Start 2021-05-31 (Actual); Primary Completion 2023-05-31 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Rate of organised colorectal cancer screening at 24 months | 24 months
  The impact of training general practitioners in motivational interviewing on the rate of organised colorectal cancer screening will be assessed by determining whether or not the immunological test proposed as part of organised colorectal cancer screening at 24 months will be carried out.

SECONDARY OUTCOMES:
Rate of organised colorectal cancer screening at 12 months | 12 months
  Whether or not to perform the proposed immunological test as part of organized colorectal cancer screening at 12 months.
Changes in perceptions of colorectal cancer screening | Day 0, 6 months, 12 months and 24 months
  Changes in perceptions of colorectal cancer screening will be assessed using a Health Belief Model (HBM). The Health Belief Model (HBM) is a social psychological health behavior change model developed to explain and predict health-related behaviors, particularly in regard to the uptake of health services.
  This Health Belief Model use for this study evaluate : individual perceptions (perceived susceptibility and severity), modifying factors (perceived threat and cues to action) and likelihood of action (perceived benefit and perception barriers and taking health action) at Day 0, Month 6, Month 12 and Month 24.
Evolution of the self-assessment of life expectancy | Day 0, 6 months, 12 months and 24 months
  Patients will answer a question to find out their self-assessment of life expectancy.
Identification of denial of the colorectal cancer screening | 24 months
  Understand why patients refuse colorectal cancer screening of by identificating et quantificating reasons why the patient did not realised the colorectal cancer screening at 24 months of follow up.

CONTACTS AND LOCATIONS:
Locations (53):
- France (53):
  - Dr ABALAIN, Brest
  - Dr HENRY, Brest
  - Dr PETTON-HILI, Brest
  - Dr DENIEL, Châteauneuf-du-Faou
  - Dr LE BOURHIS, Châteauneuf-du-Faou
  - Dr PERRIER, Clohars-Carnoët
  - Dr CHAPOIX, Crozon
  - Dr OLIVIER, Daoulas
  - Dr ATTENCOURT, Douarnenez
  - Dr KERVELLA, Douarnenez
  - Dr VELLY, Ergué-Gabéric
  - Dr BLANCHARD, Esquibien
  - Dr DESNOT, Esquibien
  - Dr VIALA, Esquibien
  - Dr DAOUDAL, Fouesnant
  - Dr LEFEVRE, Fouesnant
  - Dr MAGADUR, Fouesnant
  - Dr MUNCK, Guerlesquin
  - Dr POINOT, Guerlesquin
  - Dr LE FLOCH, Guilvinec
  - Dr LE GRIGNOU, Guissény
  - Dr PITMAN, Landivisiau
  - Dr COLLETER, Lanmeur
  - Dr CRENN-CORVEZ, Lanmeur
  - Dr BECK-ROBERT, Lanmeur
  - Dr BARAIS, Lannilis
  - Dr VERBEQUE MORVAN, Le Conquet
  - Dr TREBAOL, Le Faou
  - Dr GRALL, Le Relecq-Kerhuon
  - Dr BOUTERAON, Loperhet
  - Dr PIPET-PENIN, Moëlan-sur-Mer
  - Dr BEURTON-COURAUD, Pleyben
  - Dr LUCAS, Pleyben
  - Dr KERFRIDEN KERHOAS, Pleyber-Christ
  - Dr BAUTA, Plonévez-Porzay
  - Dr COGNEAU, Plonévez-Porzay
  - Dr GASNIER, Ploudalmézeau
  - Dr AOUDIA, Plouezoc'h
  - Dr LOPIN, Plougonven
  - Dr DROGOU, Plouhinec
  - Dr BODIN, Plounéour-Trez
  - Dr DE LA SOUDIERE, Plouzané
  - Dr PETIT, Pont-l'Abbé
  - Dr PREVOT, Pouldreuzic
  - Dr AUTRET, Quimper
  - Dr COROLLER, Quimper
  - Dr COUTURIER, Quimper
  - Dr JOLIVET COUTURE, Quimper
  - Dr KERGASTEL, Quimper
  - Dr BARCELO, Saint-Martin-des-Champs
  - Dr MONFORT, Saint-Yvi
  - Dr MAILLEUCHET, Spézet
  - Dr NICOLAS, Trégunc

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available beginning 42 months ending fifteen years following the final study report completion.
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement.

REFERENCES:
- [Derived] Aujoulat P, Le Goff D, Dany A, Robaskiewick M, Nousbaum JB, Derrienic J, Cariou M, Guillou M, Le Reste JY. Improvement of participation rate in colorectal cancer (CRC) screening by training general practitioners in motivational interviewing (AmDepCCR). Trials. 2022 Feb 14;23(1):144. doi: 10.1186/s13063-022-06056-8. PMID 35164836